CLINICAL TRIAL: NCT00142181
Title: Phase II Study of Campath-1H in Patients With Lymphoplasmacytic Lymphoma (Waldenstrom's Macroglobulinemia)
Brief Title: Phase II Study of Campath-1H Antibody to Treat Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Bayer (Industry); University of California, Los Angeles (Other); Northwestern University (Other); Arizona Oncology Associates (Network)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-079
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Lymphoplasmacytic Lymphoma; Waldenstrom's Macroglobulinemia
Keywords: Lymphoplasmacytic lymphoma; Waldenstrom's Macroglobulinemia; Antibody; Campath-1H
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab

ARMS (1):
- Campath-1H (Experimental): 30 mg IV three times a week, 6-12 weeks.
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H — Participant will receive three test doses of Campath-1H (3, 10, and 30mg). If this is tolerated then they will receive Campath-IH three times a week for 6 weeks.

SUMMARY:
The purpose of this study is to determine the safety and effects (good or bad) of Campath-1H antibody in the treatment of lymphoplasmacytic lymphoma.

DETAILED DESCRIPTION:
* Patients will receive 3 test doses of Campath-1H (3mg, 10mg, 30mg). If the patient tolerates these three test doses, then they will receive a total of 6 weeks of Campath-1H therapy three times a week.
* After the patient receives the first 6 weeks of therapy at the 30mg therapeutic dose they will be re-assessed by blood testing. If it is determined that their disease has progressed in the period of time while the patient was on Campath-1H, the patient will be removed from the study.
* If it is determined that the patient has achieved a complete remission after 6 weeks of Campath-1H treatment a bone marrow biopsy will be performed to confirm complete remission and the patient will not receive any additional treatment but will be followed for a period of 2 years.
* If the disease has remained stable or partial response has been achieved the patient will enter the second phase of therapy in which they will receive an additional 6 weeks of Campath-1H therapy. The patient will then be reassessed as described above.
* No additional therapy (as part of this study) will be performed after a 12 week course of Campath-1H.
* While the patient is on Campath-1H blood test will be performed at 3-6 month intervals over a period extending for 2 years following the last treatment. Bone marrow biopsies and/or aspirations will be conducted as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoplasmacytic lymphoma including patients with Waldenstrom's macroglobulinemia
* Adequate organ function: ANC > 500/ul; PLT > 25,000/ul; serum creatinine < 2.5; serum total bilirubin and SGOT < 2.5 times the upper normal limit.
* Age greater than 18 years
* Life expectancy of 6 months or greater
* ECOG performance status of 0-2

Exclusion Criteria:

* Chemotherapy, steroid therapy, or radiation therapy within 21 days of study entry.
* Prior Campath-1H or monoclonal antibody therapy within 3 months of study entry.
* Pregnant women
* Serious co-morbid disease, uncontrolled bacterial, fungal, or viral infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2003-03; Primary Completion 2005-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of Campath-1H in treating patients with Waldenstrom's macroglobulinemia. | 2 years

SECONDARY OUTCOMES:
To determine the safety of Campath-1H. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Isreal Deaconness Medical Center, Boston, Massachusetts
  - Dana-farber Cancer Insitiute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Treon SP, Soumerai JD, Hunter ZR, Patterson CJ, Ioakimidis L, Kahl B, Boxer M. Long-term follow-up of symptomatic patients with lymphoplasmacytic lymphoma/Waldenstrom macroglobulinemia treated with the anti-CD52 monoclonal antibody alemtuzumab. Blood. 2011 Jul 14;118(2):276-81. doi: 10.1182/blood-2011-02-338558. Epub 2011 May 12. PMID 21566092